CLINICAL TRIAL: NCT01466348
Title: Effects of a Common Cold Treatment on Cognitive Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C6930943
Record Dates: First submitted 2011-11-03; First posted 2011-11-07 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-09

CONDITIONS: Common Cold
Keywords: Paracetomol; Caffeine; Common cold
MeSH Terms: conditions — Common Cold | interventions — Acetaminophen; Caffeine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol and Caffeine (Experimental): Paracetamol and caffeine
  Interventions: Drug: Paracetamol and Caffeine
- Paracetamol (Active Comparator): Paracetamol
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol and Caffeine — Paracetamol 1000 mg and caffeine 130 mg
  Arms: Paracetamol and Caffeine
Drug: Paracetamol — Paracetamol 1000 mg
  Arms: Paracetamol

SUMMARY:
A reduction in alertness and lower levels of performance are commonly associated with the common cold. Paracetamol has been shown to be more effective than placebo in treating symptoms associated with upper respiratory tract infection; caffeine has been shown to increase levels of alertness and improve performance of people suffering from colds. This study will investigate any improvement in alertness and performance based on cognitive function and mood assessment in subjects suffering from the common cold, when taking a novel paracetamol and caffeine combination verses paracetamol alone.

ELIGIBILITY:
Inclusion Criteria:

* Present with symptoms of the common cold of no more than 96 hours duration
* Score of "2" or more on a self-rating for malaise and at least 4 other cold symptoms

Exclusion Criteria:

* Pregnancy or lactation
* Hypersensitivity to drugs
* Have taken caffeine in the last 12 hours or treated their cold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Common Cold Centre, Cardiff, Wales, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: A total of 75 participants were screened, and 72 were randomized. 3 participants did not meet the study criterion. A 5 hour washout period was maintained between treatment periods.
Groups:
- Paracetamol/ Caffeine Tablet Then Paracetamol Powder: Participants were orally administered with 200 millilitre (mL) solution of two soluble tablets, [each tablet containing 500 milligram (mg) paracetamol and 65 mg of caffeine], then 200 mL solution of paracetamol soluble powder (1000 mg). A washout period of 5 hours was maintained.
- Paracetamol Powder Then Paracetamol/ Caffeine Tablet: Participants were orally administered with 200 mL solution of paracetamol soluble powder (1000 mg), then 200 mL solution of two soluble tablets [each tablet containing 500 mg paracetamol and 65 mg of caffeine]. A washout period of 5 hours was maintained.
Period: Period I - First Intervention
Arm/Group | Paracetamol/ Caffeine Tablet Then Paracetamol Powder | Paracetamol Powder Then Paracetamol/ Caffeine Tablet
Started | 36 | 36
Intent To Treat (ITT) Population | 36 | 35 (1 participant withdrew prior receiving the treatment)
Completed | 36 | 35
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period II - Second Intervention
Arm/Group | Paracetamol/ Caffeine Tablet Then Paracetamol Powder | Paracetamol Powder Then Paracetamol/ Caffeine Tablet
Started | 35 | 36
Completed | 35 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were evaluated for baseline measures.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 71
Age Continuous [Mean (Standard Deviation); unit: Years] | 20.8 (4.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Number of Valid Responses to Rapid Visual Information Processing (RVIP) Cognitive Test
Description: The RVIP assessed the performance of visual attention mechanisms in remaining vigilant to periodically occurring events. Participants monitored a series of single numbers (0-9) appearing in the centre of the screen. During the RVIP task, participants responded to consecutive sequences of three odd or three even numbers by pressing the corresponding response button as quickly and accurately as possible. The test lasted approximately 9 minutes and mean number of valid responses to stimulus was calculated.
Time Frame: Baseline to 30 minutes post treatment administration
Population: Intent-To-Treat (ITT) population: All randomized participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Valid responses
Groups:
- Paracetamol/ Caffeine Tablet: Participants were orally administered with 200 mL solution of two soluble tablets, each tablet containing 500 mg paracetamol and 65 mg of caffeine.
- Paracetamol Powder: Participants were orally administered with 200 mL solution of 1000 mg paracetamol soluble powder.
Arm/Group | Paracetamol/ Caffeine Tablet | Paracetamol Powder
Number analyzed (Participants) | 71 | 71
Valid responses | 4.8 (0.80) | 1.3 (0.80)
Statistical Analysis 1: Comparison: Paracetamol/ Caffeine Tablet vs Paracetamol Powder; Null hypothesis was no difference in treatments in the change from baseline in the number of valid responses from the RVIP; Test type: Superiority or Other; p = 0.0008, ANOVA; No baseline covariate adjustment was carried out; Adjusted Mean Difference = 3.6, 95% CI 2-sided [1.5 to 5.6] — A positive difference favors the paracetamol/ caffeine treatment

2. Secondary Outcome: Adjusted Mean Change From Baseline in Number of Valid Responses to RVIP Cognitive Test
Description: as for outcome 1
Time Frame: Baseline to 60 minutes post treatment administration
Population: ITT population: All randomized participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Valid responses
Arm/Group | Paracetamol/ Caffeine Tablet | Paracetamol Powder
Number analyzed (Participants) | 71 | 71
Valid responses | 7.1 (0.93) | 0.6 (0.93)
Statistical Analysis 1: Comparison: Paracetamol/ Caffeine Tablet vs Paracetamol Powder; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; No baseline covariate adjustment was applied; Adjusted Mean Difference = 6.5, 95% CI 2-sided [4.5 to 8.4] — A positive difference favors the paracetamol/ caffeine treatment

3. Secondary Outcome: Adjusted Mean Change in Baseline in Valid Reaction Time to RVIP Cognitive Test
Description: The RVIP assessed the performance of visual attention mechanisms in remaining vigilant to periodically occurring events. Participants monitored a series of single numbers (0-9) appearing in the centre of the screen. During the RVIP task, participants responded to consecutive sequences of three odd or three even numbers by pressing the corresponding response button as quickly and accurately as possible. Mean valid reaction time was determined.
Time Frame: Baseline, 30 minutes and up to 60 minutes post treatment administration
Population: ITT population: All randomized participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | Paracetamol/ Caffeine Tablet | Paracetamol Powder
Number analyzed (Participants) | 71 | 71
milliseconds (msec)
  30 minutes | 6.00 (3.916) | 1.88 (3.916)
  60 minutes | 0.08 (3.983) | -4.85 (3.954)

4. Secondary Outcome: Mean Change From Baseline in Number of Incorrect and Missed Responses to RVIP Cognitive Test
Description: as for outcome 1
Time Frame: Baseline, 30 minutes and up to 60 minutes post treatment administration
Population: ITT population: All randomized participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Error); unit: Responses
Arm/Group | Paracetamol/ Caffeine Tablet | Paracetamol Powder
Number analyzed (Participants) | 71 | 71
Responses
  Incorrect responses at 30 minutes | -2.3 (1.57) | -2.7 (1.52)
  Incorrect responses at 60 minutes | -1.7 (1.93) | -2.7 (1.80)
  Missed responses at 30 minutes | -4.8 (0.69) | -1.3 (0.89)
  Missed responses at 60 minutes | -7.1 (0.90) | -0.6 (1.00)

5. Secondary Outcome: Adjusted Mean Change From Baseline in Number of Valid Responses to Sustained Attention Tasks (SAT) Cognitive Test
Description: Auditory and visual attention of participants was evaluated using a validated Sustained Attention task. For the sustained visual attention task, participants were required to respond to the letter 's' every time it appears in a continuous stream of letters presented on a screen. For the sustained auditory attention task, participants responded to the number '8' every time it appears in a continuous stream of numbers presented through headphones. Total test duration was approximately 6 minutes. Mean values of valid responses to visual and auditory tests were calculated.
Time Frame: Baseline, 30 minutes and up to 60 minutes post treatment administration
Population: ITT population: All randomized participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Error); unit: Valid responses
Arm/Group | Paracetamol/ Caffeine Tablet | Paracetamol Powder
Number analyzed (Participants) | 71 | 71
Valid responses
  30 minutes | 1.8 (0.52) | -0.5 (0.51)
  60 minutes | 1.5 (0.55) | -0.7 (0.55)

6. Secondary Outcome: Mean Change From Baseline in Number of Incorrect and Missed Responses to SAT Cognitive Test
Description: Auditory and visual attention of participants was evaluated using a validated Sustained Attention task. For the sustained visual attention task, participants were required to respond to the letter 's' every time it appears in a continuous stream of letters presented on a screen. For the sustained auditory attention task, participants responded to the number '8' every time it appears in a continuous stream of numbers presented through headphones. Total test duration was approximately 6 minutes. Mean values of incorrect and missed responses to visual and auditory tests were calculated.
Time Frame: Baseline, 30 minutes and up to 60 minutes post treatment administration
Population: ITT population: All randomized participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Error); unit: Responses
Groups:
- Paracetamol/Caffeine Tablet: Participants were orally administered with 200 mL solution of two soluble tablets, each tablet containing 500 mg paracetamol and 65 mg of caffeine.
Arm/Group | Paracetamol/Caffeine Tablet | Paracetamol Powder
Number analyzed (Participants) | 71 | 71
Responses
  Incorrect responses at 30 minutes | -2.3 (0.63) | 0.1 (0.65)
  Incorrect responses at 60 minutes | -3.6 (0.71) | 0.6 (0.72)
  Missed responses at 30 minutes | -1.8 (0.59) | 0.5 (0.44)
  Missed responses at 60 minutes | -1.5 (0.54) | 0.7 (0.55)

7. Secondary Outcome: Adjusted Mean Change From Baseline in Valid Reaction Time to SAT Cognitive Test
Description: Auditory and visual attention of participants was evaluated using a validated Sustained Attention task. For the sustained visual attention task, participants were required to respond to the letter 's' every time it appears in a continuous stream of letters presented on a screen. For the sustained auditory attention task, participants responded to the number '8' every time it appears in a continuous stream of numbers presented through headphones. Total test duration was approximately 6 minutes. Mean values of valid reaction time to visual and auditory tests were calculated.
Time Frame: Baseline, 30 minutes and up to 60 minutes post treatment administration
Population: ITT population: All randomized participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Error); unit: msec
Arm/Group | Paracetamol/ Caffeine Tablet | Paracetamol Powder
Number analyzed (Participants) | 71 | 71
msec
  30 minutes | -6.49 (2.80) | -6.18 (2.75)
  60 minutes | -10.69 (3.12) | -9.45 (3.10)

8. Secondary Outcome: Adjusted Mean Change From Baseline in Number of Valid Responses to Divided Attention Task (DAT) Cognitive Test
Description: For the DAT Cognitive test, auditory and visual stimuli were simultaneously presented and participants were asked to respond to occurrences of 's' (visual) or '8' (auditory). Total test duration was approximately 6 minutes. Mean values of valid responses to visual and auditory tests were calculated.
Time Frame: Baseline, 30 minutes and up to 60 minutes post treatment administration
Population: ITT population: All randomized participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Error); unit: Valid responses
Arm/Group | Paracetamol/ Caffeine Tablet | Paracetamol Powder
Number analyzed (Participants) | 71 | 71
Valid responses
  30 minutes | 6.8 (1.00) | 2.0 (0.99)
  60 minutes | 7.4 (1.01) | 1.9 (1.00)

9. Secondary Outcome: Adjusted Mean Change From Baseline in Valid Reaction Time to DAT Cognitive Test
Description: For the DAT Cognitive test, auditory and visual stimuli were simultaneously presented and participants were asked to respond to occurrences of 's' (visual) or '8' (auditory). Total test duration was approximately 6 minutes. Mean values of valid reaction time to visual and auditory tests were calculated.
Time Frame: Baseline, 30 minutes and up to 60 minutes post treatment administration
Population: ITT population: All randomized participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Error); unit: msec
Arm/Group | Paracetamol/ Caffeine Tablet | Paracetamol Powder
Number analyzed (Participants) | 71 | 71
msec
  30 Minutes | 1.65 (2.10) | -7.42 (2.07)
  60 minutes | -5.49 (2.44) | -12.39 (2.43)

10. Secondary Outcome: Mean Change From Baseline in Number of Incorrect and Missed Responses to DAT Cognitive Test
Description: For the DAT Cognitive test, auditory and visual stimuli were simultaneously presented and participants were asked to respond to occurrences of 's' (visual) or '8' (auditory). Total test duration was approximately 6 minutes. Mean values of incorrect and missed responses to visual and auditory tests were calculated.
Time Frame: Baseline, 30 minutes and up to 60 minutes post treatment administration
Population: ITT population: All randomized participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Error); unit: Responses
Arm/Group | Paracetamol/Caffeine Tablet | Paracetamol Powder
Number analyzed (Participants) | 71 | 71
Responses
  Incorrect responses at 30 minutes | -5.4 (0.83) | -1.4 (0.83)
  Incorrect responses at 60 minutes | -5.2 (0.77) | -0.2 (0.92)
  Missed responses at 30 minutes | -6.7 (1.19) | -2.0 (0.83)
  Missed responses at 60 minutes | -7.4 (1.24) | -1.9 (0.75)

11. Secondary Outcome: Adjusted Mean Change From Baseline in Mood Alertness and Physical Sensation Scales (MAPSS) Cognitive Test
Description: Mood patterns was evaluated using the Mood, Alertness and Physical Sensation Scales (MAPSS) which comprised of 23 questions describing moods and physical sensations, on a 9-point scale anchored at the left hand end with 'not at all' and the right hand end with 'extremely'. For each question, '9' represented the 'best' score and '1' represented the 'worst' score. Mean score was calculated by summing the responses and dividing by the number of questions answered. MAPSS Questionnaire was further divided into three main clusters: Alertness; Anxiety and Headache as per the questions.
Time Frame: Baseline, 30 minutes and up to 60 minutes post treatment administration
Population: ITT population: All randomized participants who were randomized and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Paracetamol/Caffeine Tablet | Paracetamol Powder
Number analyzed (Participants) | 71 | 71
Score on a scale
  Alertness at 30 minutes | 0.8 (0.12) | 0.2 (0.12)
  Alertness at 60 minutes | 0.7 (0.13) | 0.1 (0.13)
  Anxiety at 30 minutes | 0.2 (0.08) | 0.2 (0.08)
  Anxiety at 60 minutes | 0.3 (0.08) | 0.4 (0.08)
  Headache at 30 minutes | 0.4 (0.10) | 0.4 (0.10)
  Headache at 60 minutes | 0.6 (0.10) | 0.6 (0.10)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the start of the investigational product and until 5 days following last administration of the investigational product.
Arm/Group | Paracetamol/Caffeine Tablet | Paracetamol Powder
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71
Other Adverse Events (participants affected / at risk) | 0/71 | 0/71

LIMITATIONS AND CAVEATS:
Apparent carryover effect from the paracetamol/ caffeine treatment taken in Period 1 into the baseline assessment of Period 2 was observed, hence the statistical analysis was amended after unblinding the statistician.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.